CLINICAL TRIAL: NCT05518994
Title: Phase 2 Study to Evaluate the Clinical Efficacy and Safety of Sintilimab Plus Low-dose Bevacizumab in Patients With Astrocytoma of Different Relapse Stages
Brief Title: Sintilimab (One Anti-PD-1 Antibody) Plus Low-dose Bevacizumab for ctDNAlevel- Relapse and Clinical-relapse Astrocytoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanPPH-Astro
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: Astrocytoma of Brain
MeSH Terms: interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Subjects with ctDNA-level-relapse Astrocytoma before clinical relapse, determined according to the dynamics of TISF ctDNA.
  Interventions: Drug: Tislelizumab plus Bevacizumab
- Cohort 2 (Experimental): Subjects with clinical-relapse Astrocytoma, determined according to the response assessment in neuro-oncology (RANO) criteria for gliomas.
  Interventions: Drug: Tislelizumab plus Bevacizumab
- Cohort 3 (No Intervention): Subjects without ctDNA-level-relapse and clinical-relapse Astrocytoma.

INTERVENTIONS:
Drug: Tislelizumab plus Bevacizumab — 200mg sintilimab plus 3mg/kg bevacizumab every 3 weeks.
  Arms: Cohort 1; Cohort 2

SUMMARY:
This is an ongoing Phase 2, open-label, single-center, non-randomized study of sintilimab (one anti-PD-1 antibody same as nivolumab approved in China) plus bevacizumab administered in a low dosage schedule in adult (≥ 18 years) participants with a clinical relapse or circulating tumor DNA (ctDNA)-level relapse of Astrocytoma. This study has three non-comparative study groups. Cohort 1 and Cohort 2 will receive the same study drug sintilimab 200mg and bevacizumab 3mg/kg every 3 weeks. Cohort 3 will take only standard treatment. A stringent three-step non-randomized process will be used to assign participants to one of the study groups. Neither participants nor doctors but the researcher can choose which group participants are in. No one knows if one study group is better or worse than the other. 70 total participants are expected to participate in this study (25 participants in Cohort 1 and Cohort 2,20 participants in Cohort 3).

Grouping process: After enrollment, under the standard of care, participants will receive regular tumor in situ fluid (fluid within the surgical cavity, TISF) sampling for ctDNA analysis and recceive regular MRI. The researcher will study the TISF ctDNA and imaging dynamics to determine whether the tumor reaches to ctDNA-level (Cohort 1) or clinical relapse (Cohort 2). At the first step, all timely identified as ctDNA-level relapse tumors will be assigned into the Cohort 1 and receive the study drug immediately, those failed to be timely identified will be assigned into the Cohort 2 and receive the study drug after the clinical relapse. At the second step, once Cohort 1 or Cohort 2 reaches the target number, the new participants will be all assigned into the other Cohort. In the third step, if no ctDNA-level or clinical relapse was observed within 60 months after surgery, patients were assigned to Cohort 3 and further analyzed for prognostic biomarkers compared with Cohort 1 and Cohort 2.

DETAILED DESCRIPTION:
Primary study objectives:

-To evaluate the clinical efficacy as measured by the overall survival (OS) rate at 24 months (Cohort 2) and OS rate at 36 months (Cohort 1).

Secondary study objectives:

* To evaluate the safety/tolerability of the study treatment; To compare the OS, progression-free survival and overall response rate of the two study groups. Exploratory objectives:
* To evaluate the correlative biomarkers based on TISF ctDNA.

Standard of care:

-Surgical removal of tumors followed by adjuvant temozolomide (150-200 mg/m2, days 1-5 every 28 days for up to 12 cycles). The decision to extend TMZ treatment beyond 6 cycles, for up to 12 cycles, was left to the treating investigator. Patients were asked to attend follow-up visits every 3 months after the end of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study, including disease assessment by MRI and tumor in situ fluid (TISF) collection
3. Histologically confirmed diagnosis of Astrocytoma
4. Resection surgery done at the study center (Henan Provincial People's Hospital), with an reservoir intraoperatively implanted connecting the surgical cavity and the subscalp for postoperative noninvasive TISF collection
5. An interval of > 28 days and full recovery (i.e., no ongoing safety issues) from surgical resection prior to grouping
6. Karnofsky performance status (KPS) of 70 or higher
7. Life expectancy > 12 weeks

Exclusion Criteria:

1. More than two recurrences of Astrocytoma
2. Presence of extracranial metastatic, significant leptomeningeal disease or tumors primarily localized to the brainstem or spinal cord
3. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
4. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring chronic and systemic immunosuppressive treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects have any other condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 14 days. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalent are permitted in absence of active autoimmune disease
5. Previous radiation therapy with anything other than standard radiation therapy (i.e., focally directed radiation) administered as first line therapy
6. Previous treatment with carmustine wafer except when administered as first line treatment and at least 6 months prior to randomization
7. Previous bevacizumab or other VEGF or anti-angiogenic treatment
8. Previous treatment with a PD-1, PD-L1 or CTLA-4 targeted therapy
9. Evidence of > Grade 1 CNS hemorrhage on the baseline MRI scan
10. Inadequately controlled hypertension (defined as systolic blood pressure ≥160 mmHg and /or diastolic blood pressure ≥100 mmHg) within 7 days of first study treatment
11. Prior history of hypertensive crisis, hypertensive encephalopathy, reversible posterior leukoencephalopathy syndrome (RPLS)
12. Prior history of gastrointestinal diverticulitis, perforation, or abscess
13. Clinically significant (i.e., active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
14. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment. Any previous venous thromboembolism ≥ NCI CTCAE Grade 3 within 3 months prior to start of study treatment
15. History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month prior to randomization
16. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
17. Current or recent (within 10 days of study enrollment) use of anticoagulants that, in the opinion of the investigator, would place the subject at significant risk for bleeding. Prophylactic use of anticoagulants is allowed
18. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study
19. Minor surgical procedure (e.g., stereotactic biopsy within 7 days of first study treatment; placement of a vascular access device within 2 days of first study treatment)
20. History of intracranial abscess within 6 months prior to randomization
21. History of active gastrointestinal bleeding within 6 months prior to randomization
22. Serious, non-healing wound, active ulcer, or untreated bone fracture
23. Subjects unable (due to existent medical condition, e.g., pacemaker or ICD device) or unwilling to have a head contrast enhanced MRI
24. Positive test for hepatitis B virus surface antigen (HBV sAg) or detectable hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection
25. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
26. History of severe hypersensitivity reaction to any monoclonal antibody
27. Patients that require decadron > 4 mg/ day or equivalent of steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate at 24 months (Cohort 2) | Up to 24 months after beginning therapy
  OS-24 is the proportion of participants in the analysis population who remain alive for at least 24 months following initiation of study therapy.
Overall survival rate at 36 months (Cohort 1) | Up to 36 months after beginning therapy
  OS-36 is the proportion of participants in the analysis population who remain alive for at least 36 months following initiation of study therapy.

SECONDARY OUTCOMES:
Progression-free survival at 18 months | Up to 18 months after beginning treatment
  The proportion of participants in the analysis population who remain progression-free for at least 18 months following initiation of study therapy.
Overall survival | Up to 5 years after beginning treatment
  overall survival, as defined as time from beginning of treatment to death.
Overall response rate | Up to 5 years after beginning treatment
  Proportion of participants in the analysis population who have complete response (CR) or partial response (PR) using RANO criteria.
  Participants without efficacy evalaluation data or survival data censored at day 1. Participants without measurable disease will not be included.
Progression-free survival | Up to 5 years after beginning treatment
  Median time from allocation to first documented disease progression as per RANO or death due to any cause, whichever occurs first.
Duration of response | Up to 5 years after beginning treatment
  Time from first RANO response to disease progression in participants who achieve a PR or better.
Number of participants with treatment-emergent adverse events | Up to 5 years after beginning treatment
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) are reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, performance status evaluations, magnetic resonance imaging, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through 90 days after the last dose of durvalumab. AEs are considered to be treatment emergent if they occur or worsen in severity after the first dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xingyao Bu, Study Director — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No